CLINICAL TRIAL: NCT03771118
Title: Construction and Validation of a Simplified Provocation Test for the Diagnosis of Paracetamol Hypersensitivity
Brief Title: Drug Provocation Test (DPT) to Paracetamol
Acronym: Paracetamol
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0434
Record Dates: First submitted 2018-11-13; First posted 2018-12-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Drug Hypersensitivity
Keywords: Drug Hypersensitivity Reaction; Drug Provocation Test; Paracetamol; Reactive Doses; Reactive Times; Acetaminophen
MeSH Terms: conditions — Drug Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background : Paracetamol (acetaminophen) drug hypersensitivity reactions (DHR) are oonfirmed in about 10% of alleged cases. The diagnosis is made via an empirical drug provocation test (DPT).

Objective: Detect eliciting dose thresholds during Paracetamol DPT in order to suggest optimal step doses and to identify variables and potential risk factors associated with Paracetamol hypersensitivity.

Methods:This retrospective study, using the survival analysis and the multivariate analysis, will comprise all patients who attended the allergy service of the University Hospital of Montpellier from 1996 till 2018 with a clinical history related to Paracetamol DHR, who underwent Paracetamol DPT and who gave their consent to be included in the study. The patients are selected from the Drug Allergy & Hypersensitivity Database (DAHD).

ELIGIBILITY:
Inclusion criteria:

- Patients with a positive or negative DPT to paracetamol

Exclusion criteria:

* Patients refusing to take part in the study
* Patient under 10 years old

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient consulting in our allergy unit for a suspicion of drug hypersensitivity to Paracetamol and who underwent DPT.
Sampling Method: Non-Probability Sample
Enrollment: 498 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Detect of the reactive dose (RD) | 1 day
  The outcome measure of the RD : The dose that the patient reaches when the DPT is positive, divided by the total DPT dose for a given patient. This RD will be calculated for every patient with a positive DPT. New events (positive DPT) from one RD to another will be evaluated in number and severity.

SECONDARY OUTCOMES:
Measure is a positive DPT to paracetamol | 1 day
  Identifying clinical risk factors (Odds Ratio), using the binary logistic regression method, significantly associated with a positive Paracetamol DPT.
  Age at reaction, sex, presence of asthma and atopy, type and chronology of the initial reaction will be evaluated as potential risk factors. Risk factors of anaphylaxis during DPT will also be calculated, using the same variables.
  Potential variables to explain this measure will be introduced in a logistic model, in order to obtain crude and adjusted OR that could explain a positive DPT to paracetamol.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal DEMOLY, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No